CLINICAL TRIAL: NCT06223282
Title: Effects of Acute Resistance Exercise With Varying Training Volume and Rest Intervals Under Equal Load on Appetite Control, Food Reward, and Energy Intake: a Five-arm Crossover Randomized Controlled Trial
Brief Title: Effects of Exercise on Energy Intake-Prescription of Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202112HM039
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Eating Behavior; Food Reward
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- short inter-set rest (Experimental): 3 multi-joints resistance exercise with short (60s) inter-set rest
  Interventions: Other: short inter-set rest resistance exercise
- medium inter-set rest (Experimental): 3 multi-joints resistance exercise with medium(120s) inter-set rest
  Interventions: Other: medium inter-set rest
- long inter-set rest (Experimental): 3 multi-joints resistance exercise with long (180s) inter-set rest
  Interventions: Other: long inter-set rest
- medium inter-set rest with failure (Experimental): 3 multi-joints resistance exercise with medium (120s) inter-set rest repeated to failure each set
  Interventions: Other: medium inter-set rest with failure
- control (No Intervention): stayed sedentary during the period.

INTERVENTIONS:
Other: short inter-set rest resistance exercise — Subjects in short inter-set rest trial performed 3 sets per exercise, 7 repetitions with load of 70%-1RM with 60 sec of rest between sets.
  Arms: short inter-set rest
Other: medium inter-set rest — Subjects in medium inter-set rest trial performed 3 sets per exercise, 7 repetitions with load of 70%-1RM with 120 sec of rest between sets.
  Arms: medium inter-set rest
Other: long inter-set rest — Subjects in long inter-set rest trial performed 3 sets per exercise, 7 repetitions with load of 70%-1RM with 180 sec of rest between sets.
  Arms: long inter-set rest
Other: medium inter-set rest with failure — Subjects in long inter-set rest trial performed 3 sets per exercise, repeated to failure with load of 70%-1RM with 120 sec of rest between sets.
  Arms: medium inter-set rest with failure

SUMMARY:
Healthy young males will complete five trials in a randomized crossover counter-balanced order, including three different inter-set rest of resistance exercise in equal training volume, one repeated until failure and sedentary control. During each trial, blood samples will be collected.

The investigators hypothesized that different inter-set rest and training volume would affect subjective appetite and energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-30
* Healthy male

Exclusion Criteria:

* No acute or chronic musculoskeletal symptoms
* Smoking
* Alcohol or drug abuse
* Failure to conduct resistance exercise

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Subjective appetite | 4-hour during each study intervention
  The appetite perceptions were obtained through a 0-100 mm visual analog scale. The variables assessed included perceptions of hunger (i.e., "How hungry do you feel?"), satisfaction (i.e., "How satisfied do you feel?"), fullness (i.e., "How full do you feel?"), prospective food consumption (i.e., "How much do you think you can eat?"), and nausea (i.e., "How nauseous do you feel?"), with 0 indicating "not at all" and 100 signifying "extremely.".
Change in acyl-Ghrelin | 4-hour during each study intervention
  acyl-Ghrelin in pg/mL
Change in total-Ghrelin | 4-hour during each study intervention
  total-Ghrelin in pg/mL
Change in PYY | 4-hour during each study intervention
  PYY in pg/mL
Change in active-GLP-1 | 4-hour during each study intervention
  active-GLP-1 in pg/mL
Change in total-GLP-1 | 4-hour during each study intervention
  total-GLP-1 in pg/mL
Change in lactate | 4-hour during each study intervention
  insulin in mmol/L

SECONDARY OUTCOMES:
Explicit liking | 4 hours during each study intervention
  A visual analog scale ranging from 0 to 100 mm was utilized to evaluate the question, "How pleasant would it be to taste some of this food now?" with 0 indicating "not at all" and 100 signifying "extremely."
Explicit wanting | 4 hours during each study intervention
  A visual analog scale ranging from 0 to 100 mm was utilized to evaluate the question, "How much do you want some of this food now?" with 0 indicating "not at all" and 100 signifying "extremely."
Implicit wanting | 4 hours during each study intervention
  Participants were given a set of food image pairs and were asked to select their preference by answering the question, "Which food do you desire the most at the moment?". The implicit wanting calculation involved further consideration of response time data based on preference choices using a standardized equation.
Relative preference | 4 hours during each study intervention
  Participants were given a set of food image pairs and were asked to select their preference by answering the question, "Which food do you desire the most at the moment?". The relative preference was the sum of the times each type of food was chosen, with a maximum value of 48 and a minimum value of 0.
Fat appeal bias | 4 hours during each study intervention
  Fat preference (high or low) was calculated by subtracting the mean low-fat scores from the mean high-fat scores. Positive values suggest a preference for high-fat foods, while negative scores indicate a preference for low-fat or savory foods, and a score of 0 signifies an equal preference between fat content.
Taste appeal bias | 4 hours during each study intervention
  Taste preference (savoury or sweet) was calculated by subtracting the mean savory scores from the mean sweet scores. Positive values suggest a preference for sweet foods, while negative scores indicate a preference for savory foods, and a score of 0 signifies an equal preference between taste categories.
Change in glucose | 4 hours during each study intervention
  glucose in mg/dL
Change in TG | 4 hours during each study intervention
  TG in mg/dL
Change in insulin | 4 hours during each study intervention
  insulin in mU/L
Energy intake | 3 days during each study intervention
  Participants are required to record their diet for the day before, the current day, and the day following the experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Wen Liu, Ph.D., Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan